CLINICAL TRIAL: NCT02487537
Title: Immediate and Long-term Induction of Incretin Release by Artificial Sweeteners 2
Acronym: ILIAS-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: German Institute of Human Nutrition (Other)
Collaborators: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. Andreas F. H. Pfeiffer, Director, Department of Clinical Nutrition, German Institute of Human Nutrition
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: ILIAS-2
Record Dates: First submitted 2015-03-23; First posted 2015-07-01 (Estimated); Last update posted 2020-06-24 (Actual); Status verified 2020-06

CONDITIONS: Diabetes; Pre-diabetes
Keywords: incretin release
MeSH Terms: conditions — Diabetes Mellitus; Glucose Intolerance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Non-sweetened soft drink (Placebo Comparator): 4-week-intervention with one liter of custom-made soft drink per day; soft drink does not contain glucose or any kind of sweet tasting substance
  Interventions: Dietary Supplement: custom-made soft drink
- Sweetened soft drink (Active Comparator): 4-week-intervention with one liter of custom-made soft drink per day, soft drinks contains an amount of sweetener, which is isosweet compared to 100 g of sucrose in one liter of beverage
  Interventions: Dietary Supplement: custom-made soft drink

INTERVENTIONS:
Dietary Supplement: custom-made soft drink

SUMMARY:
Epidemiological data suggest, that not only sugar-based, but also artificially sweetened soft drinks may play a role in the development of diabetes.

Recent studies in animals and humans have shown, that artificial sweeteners (AS) influence metabolic responses after glucose ingestion, possibly alter the intestinal microbiome and even modulate incretin release.

Data on human subjects are sparse and controversial, especially in a long-term manner. We therefore conduct a cross-over study to assess metabolic response to sweetened vs. non-sweetened soft drinks, which are consumed over a period of 4 weeks.

DETAILED DESCRIPTION:
Epidemiological data suggest, that not only sugar-based, but also artificially sweetened soft drinks may play a role in the development of diabetes.

Recent studies in animals and humans have shown, that artificial sweeteners (AS) influence metabolic responses after glucose ingestion, possibly alter the intestinal microbiome and even modulate incretin release.

Data on human subjects are sparse and controversial, especially in a long-term manner. We therefore conduct a cross-over study to assess metabolic response to sweetened vs. non-sweetened soft drinks, which are consumed over a period of 4 weeks. Metabolic assessment will be based on oral glucose tolerance tests.

ELIGIBILITY:
Inclusion Criteria:

* healthy

Exclusion Criteria:

* no metabolic disorders such as diabetes, hypothyroidism, corticoid therapy, heart or lung disease

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
change in release of GIP | 4 weeks (cross-over)
  change in fasting state and post-glucose release of GIP between the two interventions
change in release of GLP-1 | 4 weeks (cross-over)
  change in fasting state and post-glucose release of GLP-1 between the two interventions
change in release of GLP-2 | 4 weeks (cross-over)
  change in fasting state and post-glucose release of GLP-2 between the two interventions
change in release of PYY | 4 weeks (cross-over)
  change in fasting state and post-glucose release of PYY between the two interventions
change in release of insulin | 4 weeks (cross-over)
  change in fasting state and post-glucose release of insulin between the two interventions
change in combined levels of glucose and insulin, expressed in calculated indices for insulin secretion | 4 weeks (cross-over)
  change in fasting state and post-glucose insulin secretion between the two interventions
change in combined levels of glucose and insulin, expressed in calculated indices for insulin sensitivity | 4 weeks (cross-over)
  change in fasting state and post-glucose insulin sensitivity between the two interventions

CONTACTS AND LOCATIONS:
Locations (1):
- German Institut for Human Nutrition; Department for Clinical Nutrition, Bergholz-Rehbrücke, Brandenburg, Germany

REFERENCES:
- [Derived] Lohner S, Kuellenberg de Gaudry D, Toews I, Ferenci T, Meerpohl JJ. Non-nutritive sweeteners for diabetes mellitus. Cochrane Database Syst Rev. 2020 May 25;5(5):CD012885. doi: 10.1002/14651858.CD012885.pub2. PMID 32449201